CLINICAL TRIAL: NCT02956681
Title: Statewide Communication to Reach Diverse Low Income Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Prevention Institute of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSF-SW-2007; R01CA129096 (NIH)
Record Dates: First submitted 2016-05-17; First posted 2016-11-07 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed Intervention Group (Active Comparator): In this arm of the randomized delayed intervention control trial, participants randomized to delayed intervention control group were sent a brochure with information on hereditary breast and ovarian cancer and the phone number to call a cancer risk program for free genetic counseling.
  Interventions: Behavioral: Delayed Intervention Group
- Intervention Group (Active Comparator): In this arm of the randomized delayed intervention control trial, those randomized to the intervention group were told that because of their family history, we were able to offer them a free genetic counseling appointment.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Callers to California's toll-free breast/cervical screening phone service were screened for family history. Callers identified as high risk will be told that a genetic counselor will call them back to offer them a free genetic counseling appointment and that a brochure will be sent. A UCSF/SFGH genetic counseling assistant will call them back within a few days to offer them a free genetic counseling appointment at SFGH.
  Arms: Intervention Group
Behavioral: Delayed Intervention Group — This is a randomized delayed intervention control trial in which eligible callers to California's toll-free breast/cervical screening phone service were screened for family history. Callers identified as high risk will be told that they are eligible to speak to a genetic counselor who is available at no charge at SFGH and that they will be sent a brochure with information on where to call.
  Arms: Delayed Intervention Group

SUMMARY:
Recruitment for prevention, and early detection among health disparities populations represents a major challenge in chronic disease control. This effect is magnified for individuals at high risk for conditions such as genetic breast cancer or chronic hepatitis. Costs are typically high, particularly given the common practice of developing a single outreach channel to address each disease or condition. In a randomized delayed intervention control trial, the investigators tested a strategy to identify low-income women at high risk for hereditary breast and ovarian cancer (HBOC) outside the clinical setting and refer them to free genetic counseling.

DETAILED DESCRIPTION:
This study addresses a disparity in services related to the rare but serious condition of HBOC. In a randomized delayed intervention control trial, the investigators were able to identify high-risk but predominantly unaffected women among callers seeking referrals to free cancer screening. The investigators compared an immediate offer of a genetic counseling appointment to information on hereditary breast and ovarian cancer sent by mail. Our study demonstrated that when a diverse population of low-income women calls a trusted information and referral source, it is possible to both engage them on a topic that is different from the purpose for their call and to recruit them for participation in research.

Our intervention was designed to fit as seamlessly as possible with two end user organizations. Existing staff (Information Specialists) of the state's phone service administered a simple family history screener similar to their usual procedure for assessing eligibility for free mammography. Cancer Risk Program Genetic Counseling Assistants followed up with an outcall, just as they do normally in response to family history screeners filled out in the hospital's mammography clinic. Our results not only showed a significantly larger effect on use of genetic counseling with the call and appointment offer compared with a mailed brochure, it was clear from calls made to women in both arms after the intervention period that calling is not only effective but essential to encourage use of genetic counseling in this population. The number of women counseled in the intervention group was initially much higher than the control group, and additional intervention group members obtained counseling when called again after the two month intervention period. The addition of genetic counseling by phone enabled a substantial number of women to obtain counseling who would not have done so otherwise. Our study demonstrated that, for the complex and highly personal issue of HBOC, multiple attempts over a period of months are needed and justified.

ELIGIBILITY:
Inclusion Criteria

* Residence within one of six local counties (for ease of access to our sites offering free genetic counseling and testing), age 25+, and English- or Spanish-speaking (the languages in which genetic counseling was conducted at risk program sites).

Exclusion Criteria

* American Indian/Alaska Native and Native Hawaiian/Other Pacific Islander will not be included since very few call EWC.
* Children (individuals under 25 years of age) will not be included in the study.
* The rationale for this exclusion is that the research topic is not relevant to children.
* The EWC does not target children, whose medical care is typically under the control of their parents or guardians.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Receipt of Genetic Counseling During Intervention Period | Up to three years
  The primary outcome measure is receipt of genetic counseling within the two month intervention period.

SECONDARY OUTCOMES:
Time to Counseling | Up to three years
  The study arms were compared with respect to time from randomization to counseling appointment using the log-rank test, and Kaplan-Meier curves were computed for each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Rena J Pasick, DrPH, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No